CLINICAL TRIAL: NCT05819008
Title: Remote Neuropsychological Assessment of Patients With Neurological Disorders and Injuries
Status: Recruiting | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Nils Berginström, Associate Professor, Umeå University
Other Study IDs: 7004076
Record Dates: First submitted 2023-03-21; First posted 2023-04-19 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury; Stroke; Multiple Sclerosis; Parkinson Disease; Epilepsy; Brain Tumor
Keywords: Neuropsychological assessment
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Multiple Sclerosis; Parkinson Disease; Epilepsy; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with neurological disorders or injuries and Healthy Controls
  Interventions: Diagnostic Test: Neuropsychological Assessment

INTERVENTIONS:
Diagnostic Test: Neuropsychological Assessment — To validate Mindmore Distance (MD), the following standard neuropsychological tests will be used in a testing session with a psychologist:
  * Wordlist 1 and 2 from WMS-III (Wechsler, 1997). Equivalent to RAVLT in MD
  * Coding from WAIS-IV (Wechsler, 2008). Equivalent to SDPT in MD
  * Block Span from WMS-III (Wechsler, 1997). Equivalent to CBT in MD
  * Trail Making Test from D-KEFS (Delis et al., 2001). Equivalent to TMT-Click in MD
  * Color-Word Interference Test from D-KEFS. Equivalent to Stroop in MD
  * Verbal fluency from D-KEFS. Equivalent to FAS in MD
  All participants will complete some questionnaires: Hospital Anxiety and Depression Scale (Zigmond & Snaith, 1983); Insomnia Severity Index (Bastien, Vallieres, & Morin, 2001); Cognitive Failure Questionnaire (Broadbent, Cooper, FitzGerald, & Parkes, 1982); Perceived Stress Scale (Levenstein et al., 1993); Multidimensional Fatigue Inventory (Smets, Garssen, Bonke, & De Haes, 1995).

SUMMARY:
For the last decades, many aspects of human life have been altered by digital technology. For health care, this have opened a possibility for patients who have difficulties travelling a long distance to a hospital to meet with their health care providers over different digital platforms. With an increased digital literacy, and an aging population often living in the countryside, far from hospitals or other health care settings, an increasing need for digitalization of meetings between patients and health care personnel is inevitable.

However, neuropsychological assessment is one sort of health care not possible to directly transfer into digital form. These evaluations are most often performed with well validated tests, only to be used in a paper-pencil form with a specially trained psychologist during physical meetings.

The aim of this project is to investigate whether a newly developed digital neuropsychological test battery can be used to perform remote assessments of cognitive function in patients with neurological injuries and impairments. To this date, there are no such test batteries available in the Swedish language.

Mindmore (www.mindmore.com) is a test system developed in Sweden, performing neuropsychological tests on a tablet, but still with the psychologist present in the room. This system is now evolving into offering the possibility for the patient to perform the test in their own home, using their own computer or tablet. The aim of the present research project is to validate this latter system (Mindmore Distance), using the following research questions:

1. Are the tests in Mindmore Distance equivalent to traditional neuropsychological tests in patients with traumatic brain injury, stroke, multiple sclerosis, Parkinson's Disease, epilepsy, and brain tumor?
2. Can the results from Mindmore Distance be transferred into neuropsychological profiles that can be used in diagnostics for specific patient groups?
3. How do the patients experience undergoing a neuropsychological evaluation on their own compared to traditional neuropsychological assessment in a physical meeting with a psychologist?

DETAILED DESCRIPTION:
The neurological disorders and injuries are characterized by damage to neurons in the central nervous system. Since many of these damages affect the brain, rudimentary functions of the brain, including cognition, are often affected in these patient groups which include traumatic brain injuries, stroke, multiple sclerosis, Parkinson's Disease, epilepsy and different forms of brain tumors.

Neuropsychological assessment of cognitive functions plays a central role in both diagnostics and evaluation as well as planning of treatment and rehabilitation for these patients. Today, the neuropsychological evaluation is often used as an objective way of determining cognitive dysfunction that can be used for medical statements about ability to work, or to establish level of functioning in insurance cases.

Traditional neuropsychological assessment is performed in a physical meeting between the patient and a psychologist in charge of the examination, where different cognitive functions are assessed. For example, the psychologist can read out loud words or numbers to be remembered by the patient (working and long-term memory), the patient might search for a specific target on a piece of paper (attention or mental speed), or that the patient is instructed to say as many words as possible starting with a specific letter (verbal fluency and executive functions). The same function is often tested with different tests to validate the results, and the results are interpreted in the light of the patient's behavior and amnestic information. After the testing session, the psychologist is faced with an often time-demanding task of scoring and comparing the results to normative data. Since the start of the new millennium, computer-based tests or a combination of computers and "paper-pencil tests" of tablets have become more common in clinical use. These have reduced some the time that the psychologist has to spend on scoring, but still mean that the patient has to come to the clinic to undergo the neuropsychological examination.

During the corona pandemic, many health care visits were cancelled, when many patients, especially in the older population, had to minimize the risk of infection. In Sweden, a large and sparsely populated country, another challenge to physical meetings in health care is long and demanding travels for patients. Thus, many visits to health care, both before and during the pandemic, has be transferred to digital form and online platforms.

Neuropsychological evaluations are however not directly transferable into digital form. Both reliability and validity of the neuropsychological assessment are highly reliant on standardization of instructions and administration procedures. Since the results from the tests are compared to the results of a normal population, where the standardized administration procedure has been used, it is very important that the testing with patients are performed in the same way. If the administration procedure is changed too much, the results will not be reliable nor valid. Systematic reviews and meta analyses have shown that some verbal tests may be possible to perform in a video conference meeting, but for tests involving motor or visual processing, this cannot be recommended.

Thus, there is a need for the development of instruments that can enable psychologists to perform neuropsychological evaluations remotely, where both administration and scoring are performed automatically, saving cost and time for the health care system. Mindmore (www.mindmore.com) is a digital neuropsychological test battery developed in Sweden and it has been validated in a Swedish healthy population, and normative data has been collected. Included in this battery are tests of audioverbal learning and episodic memory, mental speed, working memory and executive functions in the form of inhibition, shifting and verbal fluency. However, this system still requires a visit to health care where the testing is performed. Now, Mindmore is launching a self-administered desktop version of this battery, Mindmore Distance, which can be performed on any computer or tablet with an internet connection. This is the first Swedish test on the market able to perform neuropsychological tests remotely. It is very important that neuropsychological tests are developed, validated and normed in the countries where they will be used clinically, since language, culture and education affect results on these tests at a very high degree. Mindmore Distance is right now being validated and normed in a healthy Swedish population, but no study has been performed on patients. Validating test in specific patient groups is critical since this can answer whether the tests are suitable for the patients and to see if the tests are possible to use to discriminate between different patient groups or between patients and healthy controls.

In a cross-sectional design, patients with neurological disorders or injuries will be tested using Mindmore Distance at home, and traditional neuropsychological test with a neuropsychologist at Neuro-Head-Neck-Centre (NHHC) at the Umeå University Hospital, Umeå, Sweden. Patient groups included are: Traumatic brain injury (TBI), Stroke, Multiple sclerosis, Parkinson's Disease, Epilepsy and Brain Tumors.

When referred to neuropsychological examination at NHHC, patients will receive written information about the project and contact information to the principal investigator to whom they can turn for questions. If they wish to participate, a link in the letter will take them to the research person information, where they can sign informed consent using Scrive e-sign (scrive.com) and digital identification (BankID). After this, patients will be randomized to performing standard neuropsychological assessment at the clinic or Mindmore Distance at home first. This randomization procedure is used to control for test-retest or learning effects.

Healthy controls will be recruited through advertising, where they through a link will reach the same page as patients. After signing informed consent, a similar randomization procedure as for patients will take place. Healthy controls will perform the physical neuropsychological examination at a specific occasion in the facilities of the Department of Psychology, Umeå University. In the same session as the traditional neuropsychological evaluation, both patients and healthy controls will complete questionnaires on demographical and health related factors.

The validity of Mindmore test will be validated against traditional paper-pencil neuropsychological test using Pearson and/or Spearman correlation coefficients, interpreted using Cohens (1992) cutoffs of weak (0.1), medium (0.3) and strong (0.5) correlations. Further, multiple linear regressions will be performed to investigate and adjust for background variables.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* Diagnosed with a neurological disorder or injury, alternatively under medical examination for such a diagnosis
* Owns and can handle a computer with internet connection

Exclusion Criteria:

* Severe psychiatric disorder, such a schizophrenia, severe depression
* Addiction of alcohol or other substances
* Not speaker of Swedish
* On sedatives, such as sleep or pain medication
* Multiple neurological diagnoses
* Not being able to participate in a neuropsychological examination, or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients treated at the Neuro-Head-Neck-Center (NHHC) at Umeå University hospital. When referred to neuropsychological examination at NHHC, patients will receive written information about the project and contact information to the principal investigator to whom they can turn for questions, before signing informed consent.
  Patient groups included are:
  * Traumatic brain injury (TBI), including patients with persisting symptoms after concussion, post-concussional disorder.
  * Stroke
  * Multiple sclerosis
  * Parkinson's Disease
  * Epilepsy
  * Brain Tumors
  A comparison group of healthy volunteers will be recruited using advertising.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Validity of Rey Auditory Verbal Learning Test in Mindmore | Baseline
  The results of RAVLT in Mindmore will be validated against Word List Recall from Wechsler Memory Scale - Third edition.
Validity of Symbol Digit Processing Test in Mindmore | Baseline
  The results of SDPT in Mindmore will be validated against Coding from Wechsler Adult Intelligence Scale - Fourth edition.
Validity of Corsi Block Test in Mindmore | Baseline
  The results of CBT in Mindmore will be validated against Block Span from Wechsler Memory Scale - Third edition.
Validity of Trail Making Test - Click in Mindmore | Baseline
  The results of TMT-Click in Mindmore will be validated against Trail Making Test from Delis-Kaplan Executive Functions System.
Validity of Stroop in Mindmore | Baseline
  The results of Stroop in Mindmore will be validated against Color-Word Interference Test from Delis-Kaplan Executive Functions System.
Validity of FAS in Mindmore | Baseline
  The results of FAS in Mindmore will be validated against Verbal Fluency from Delis-Kaplan Executive Functions System.

CONTACTS AND LOCATIONS:
Overall Officials: Nils Berginström, PhD, Principal Investigator — Umeå Universitet, Department of Psychology
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Benedict RHB, Amato MP, DeLuca J, Geurts JJG. Cognitive impairment in multiple sclerosis: clinical management, MRI, and therapeutic avenues. Lancet Neurol. 2020 Oct;19(10):860-871. doi: 10.1016/S1474-4422(20)30277-5. Epub 2020 Sep 16. PMID 32949546
- [Background] Bjorngrim S, van den Hurk W, Betancort M, Machado A, Lindau M. Comparing Traditional and Digitized Cognitive Tests Used in Standard Clinical Evaluation - A Study of the Digital Application Minnemera. Front Psychol. 2019 Oct 18;10:2327. doi: 10.3389/fpsyg.2019.02327. eCollection 2019. PMID 31681117
- [Background] Brearly TW, Shura RD, Martindale SL, Lazowski RA, Luxton DD, Shenal BV, Rowland JA. Neuropsychological Test Administration by Videoconference: A Systematic Review and Meta-Analysis. Neuropsychol Rev. 2017 Jun;27(2):174-186. doi: 10.1007/s11065-017-9349-1. Epub 2017 Jun 16. PMID 28623461
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Buckley RF, Sparks KP, Papp KV, Dekhtyar M, Martin C, Burnham S, Sperling RA, Rentz DM. Computerized Cognitive Testing for Use in Clinical Trials: A Comparison of the NIH Toolbox and Cogstate C3 Batteries. J Prev Alzheimers Dis. 2017;4(1):3-11. doi: 10.14283/jpad.2017.1. PMID 29188853
- [Background] Daniel MH, Wahlstrom D, Zhang O. Equivalence of Q-interactive® and Paper Administrations of Cognitive Tasks: WISC®-V. NCS Pearson Inc.; 2014.
- [Background] Delis DC, Kaplan E, Kramer JH. D-KEFS - Delis Kaplan Executive Functions System - Technical Manual. San Antonio: Pearson; 2001.
- [Background] Dikmen SS, Machamer JE, Winn HR, Temkin NR. Neuropsychological Outcome at 1-Year Post Head-Injury. Neuropsychology. 1995;9(1):80-90.
- [Background] van der Naalt J, van Zomeren AH, Sluiter WJ, Minderhoud JM. One year outcome in mild to moderate head injury: the predictive value of acute injury characteristics related to complaints and return to work. J Neurol Neurosurg Psychiatry. 1999 Feb;66(2):207-13. doi: 10.1136/jnnp.66.2.207. PMID 10071101
- [Background] Sun JH, Tan L, Yu JT. Post-stroke cognitive impairment: epidemiology, mechanisms and management. Ann Transl Med. 2014 Aug;2(8):80. doi: 10.3978/j.issn.2305-5839.2014.08.05. PMID 25333055
- [Background] Yang Y, Tang BS, Guo JF. Parkinson's Disease and Cognitive Impairment. Parkinsons Dis. 2016;2016:6734678. doi: 10.1155/2016/6734678. Epub 2016 Dec 12. PMID 28058128
- [Background] Holmes GL. Cognitive impairment in epilepsy: the role of network abnormalities. Epileptic Disord. 2015 Jun;17(2):101-16. doi: 10.1684/epd.2015.0739. PMID 25905906
- [Background] Pendergrass JC, Targum SD, Harrison JE. Cognitive Impairment Associated with Cancer: A Brief Review. Innov Clin Neurosci. 2018 Feb 1;15(1-2):36-44. PMID 29497579
- [Background] Lezak MD, Howieson DB, Loring DW. Neuropsychological Assessment. 4 ed. New York: Oxford University Press; 2004.
- [Background] Germine L, Reinecke K, Chaytor NS. Digital neuropsychology: Challenges and opportunities at the intersection of science and software. Clin Neuropsychol. 2019 Feb;33(2):271-286. doi: 10.1080/13854046.2018.1535662. Epub 2019 Jan 6. PMID 30614374
- [Background] Vermeent S, Dotsch R, Schmand B, Klaming L, Miller JB, van Elswijk G. Evidence of Validity for a Newly Developed Digital Cognitive Test Battery. Front Psychol. 2020 Apr 24;11:770. doi: 10.3389/fpsyg.2020.00770. eCollection 2020. PMID 32390918
- [Background] Wechsler D. Wechsler Adult Intelligence Scale-Fourth Edition. San Antonio: Pearson; 2008.
- [Background] Marra DE, Hamlet KM, Bauer RM, Bowers D. Validity of teleneuropsychology for older adults in response to COVID-19: A systematic and critical review. Clin Neuropsychol. 2020 Oct-Nov;34(7-8):1411-1452. doi: 10.1080/13854046.2020.1769192. Epub 2020 Jun 10. PMID 32519594
- [Background] van den Hurk W, Bergman I, Machado A, Bjermo J, Gustavsson A. Swedish Normative Data for Mindmore: A Comprehensive Cognitive Screening Battery, Both Digital and Self-Administrated. J Int Neuropsychol Soc. 2022 Feb;28(2):188-202. doi: 10.1017/S135561772100045X. Epub 2021 May 24. PMID 34027854
- [Background] Ardila A. Directions of research in cross-cultural neuropsychology. J Clin Exp Neuropsychol. 1995 Feb;17(1):143-50. doi: 10.1080/13803399508406589. PMID 7608296
- [Background] Mitrushina MN, Boone KB, D'Elia LF. Handbook of Normative Data for Neuropsychological Assessment. New York: Oxford University Press; 1999.
- [Background] Wechsler D. Wechsler Memory Scale - Third Edition. San Antonio: Psychological Corporation; 1997.
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Levenstein S, Prantera C, Varvo V, Scribano ML, Berto E, Luzi C, Andreoli A. Development of the Perceived Stress Questionnaire: a new tool for psychosomatic research. J Psychosom Res. 1993 Jan;37(1):19-32. doi: 10.1016/0022-3999(93)90120-5. PMID 8421257
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Cohen J. A power primer. Psychol Bull. 1992 Jul;112(1):155-9. doi: 10.1037//0033-2909.112.1.155. PMID 19565683
- [Derived] Berginstrom N, Andersson L. Remote neuropsychological assessment of patients with neurological disorders and injuries-a study protocol for a cross-sectional case-control validation study. BMJ Open. 2024 Apr 22;14(4):e080628. doi: 10.1136/bmjopen-2023-080628. PMID 38653513